CLINICAL TRIAL: NCT02233036
Title: Evaluating the Transition From Pediatric to Adult Care Among Adolescents With Chronic Granulomatous Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914088; 14-I-N088
Record Dates: First submitted 2014-09-04; First posted 2014-09-08 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2017-01-10

CONDITIONS: CGD
Keywords: Young Adults; Transfer; Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Background:

People who get chronic illnesses as children are living longer. When they turn 18, they switch from pediatric care to adult care. This can be a difficult change. Chronic Granulomatous Disease (CGD) is an inherited disease. It causes long-term, repeated infections. People with CGD are usually diagnosed when they are very young children. Researchers want to find out more about how young people with CGD handle the change to adult care. What they learn may make this easier for people with CGD in the future.

Objective:

- To identify what helped or hurt young adults with CGD as they went from pediatric to adult care.

Eligibility:

- Adults with CGD who were 18 24 years old between January 2011 and February 2014.

Design:

* Participants will already be enrolled in NIH studies.
* Eligible people will get materials in the mail. They will get a letter with study information, an interview questionnaire, and an information sheet.
* Researchers will call participants 1 week after the packets are sent. They will talk about the study and find out if the person wants to join.
* An interview will be completed immediately or scheduled for the future. The interview will take about 45 minutes. The researcher will ask the participant about their disease. They will also ask about travel to NIH, being an outpatient or inpatient there, and legal documents.
* Researchers may contact the subjects again by phone if they need more information at any point during the study.

DETAILED DESCRIPTION:
Children with chronic illnesses are thriving well into adulthood due to ongoing medical advances. Many healthy and typically developing 18-year-olds should be able to manage a transition from pediatric to adult care, but this transition can be challenging for adolescents with chronic illness. A poor transition to adult care can result in medical, social and educational issues for patients, families and the medical team. At issue are questions of independence and self-management: are young adult patients prepared to travel to NIH alone? Are they prepared to speak with physicians about their disease process and medications? Are they ready to give informed consent for studies in which they have been participating?

The National Institute of Allergy and Infectious Diseases (NIAID) at the National Institutes of Health (NIH) has several hundred adolescents enrolled in clinical trials, many of whom rely on NIH providers for specialized care. No formal program exists to assist these patients in the transition from pediatric to adult care. Pediatric inpatients are admitted to the adult inpatient unit when they turn 18 with little knowledge of the policy differences between the units.

The investigators propose a retrospective exploratory descriptive study to (a) identify and describe experiences that young adults found to enable or hinder their transition and (b) explore these patients ideas for enhancing the transition process. A semi-structured questionnaire administered by phone or face to face to approximately 40 young adults with chronic granulomatous disease (CGD) will gather qualitative and quantitative information about the use of inpatient and outpatient services at the NIH Clinical Center prior to and since the subjects 18th birthdays. Data will be used to develop a program to help NIAID pediatric patients with CGD transition successfully to adult care.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. 18 to 24 years of age during January 1, 2011 to December 31, 2012
2. Documented diagnosis of CGD
3. Enrolled in one of the following three NIAID protocols that investigate CGD (and other immunodeficiencies):

   * Detection and Characterization of Host Defense Defects (93-I-0119), PI: Dr. Steven Holland
   * Screening and Baseline Assessment of Patients with Abnormalities of Immune Function (05-I-0213), PI: Dr. Harry Malech
   * Screening Protocol for Detection and Characterization of Infections and Infection (07-I-0033), PI: Dr. Steven Holland
4. Record of a visit to NIH prior to 18th birthday and at least one visit during January 1, 2011 to December 31, 2012
5. Health status sufficient to participate in an interview, as determined by patient self-report at the start of the interview.
6. Fluency in English

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-03-26; Primary Completion 2016-01-11 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Successful transition to adult care | After completion of interview

SECONDARY OUTCOMES:
To explore strategies that young adult patients believe mayenhance the process of transition from pediatric to adult care | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Patricia R Driscoll, R.N., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), 9000 Rockville Pi, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fernandes SM, Landzberg MJ. Transitioning the young adult with congenital heart disease for life-long medical care. Pediatr Clin North Am. 2004 Dec;51(6):1739-48, xi. doi: 10.1016/j.pcl.2004.07.006. PMID 15561183
- [Background] Kennedy A, Sloman F, Douglass JA, Sawyer SM. Young people with chronic illness: the approach to transition. Intern Med J. 2007 Aug;37(8):555-60. doi: 10.1111/j.1445-5994.2007.01440.x. PMID 17640188
- [Background] Sawicki GS, Lukens-Bull K, Yin X, Demars N, Huang IC, Livingood W, Reiss J, Wood D. Measuring the transition readiness of youth with special healthcare needs: validation of the TRAQ--Transition Readiness Assessment Questionnaire. J Pediatr Psychol. 2011 Mar;36(2):160-71. doi: 10.1093/jpepsy/jsp128. Epub 2009 Dec 29. PMID 20040605